CLINICAL TRIAL: NCT06988124
Title: Intravenous Dexamethasone Palmitate for Prophylaxis of Postoperative Nausea and Vomiting After Craniotomy
Brief Title: Dexamethasone Palmitate for PONV After Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2025-041-02-03
Record Dates: First submitted 2025-05-13; First posted 2025-05-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — dexamethasone 21-palmitate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone palmitate group (Experimental)
  Interventions: Drug: Dexamethasone Palmitate
- Dexamethasone group (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone Palmitate — Patients in the dexamethasone palmitate group will be assigned to receive intravenous injection of dexamethasone palmitate 8 mg (contains 5mg dexamethasone) after anesthesia induction and before surgical incision.
  Arms: Dexamethasone palmitate group
Drug: Dexamethasone — Patients in the dexamethasone group will be assigned to receive intravenous injections of dexamethasone 5 mg after anesthesia induction and before surgical incision.
  Arms: Dexamethasone group

SUMMARY:
Dexamethasone is almost one of the most commonly used drugs for postoperative nausea and vomiting (PONV) prevention. However, PONV is still a complex problem to be solved; for example, even with preoperative dexamethasone administration, there are still some patients undergoing craniotomy still experience PONV within 24 hours postoperatively. Compared to dexamethasone, dexamethasone palmitate has a long-lasting anti-inflammatory effect, 2-5 times that of traditional water-soluble dexamethasone, with fewer adverse effects. This trial aims to assess the effect and safety of preoperative dexamethasone palmitate on PONV after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years;
* Providing written informed consent;
* Perform elective craniotomy undergoing general anesthesia.

Exclusion Criteria:

* Known to be allergic to dexamethasone;
* Any systemic glucocorticoids within 3 months before trial entry;
* History of severe heart disease, liver/kidney failure, or systemic rheumatic diseases (rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, et al);
* Cognitive impairment or severe mental illness;
* Uncontrolled diabetes or infectious diseases;
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of PONV | Within the first 24 hours postoperatively
  PONV will be defined as any nausea, emetic episodes (vomiting or retching), or both. Nausea is defined as an unpleasant sensation with an urge to vomit. Vomiting is defined as the physical event of forcefully expelling gastric contents through the mouth. Retching refers to the forced movement of gastrointestinal contents without actual expulsion of vomitus.

SECONDARY OUTCOMES:
The Incidence of PONV | At 6 hours, 48 hours, and 72 hours postoperatively
  PONV will be defined as any nausea, emetic episodes (vomiting or retching), or both. Nausea is defined as an unpleasant sensation with an urge to vomit. Vomiting is defined as the physical event of forcefully expelling gastric contents through the mouth. Retching refers to the forced movement of gastrointestinal contents without actual expulsion of vomitus.
Incidence of postoperative nausea (PON) and postoperative vomiting (POV) | At 6 hours, 24 hours, 48 hours, and 72 hours postoperatively
  Incidence of postoperative nausea (PON) and postoperative vomiting (POV)
The number of vomiting or retching episodes | Within 6 hours, 24 hours, 48 hours, and 72 hours postoperatively
  The number of vomiting or retching episodes
The severity of PONV | At 6 hours, 24 hours, 48 hours, and 72 hours postoperatively
  The severity of PONV will be measured using the simplified PONV impact scoring system. The simplified PONV impact scoring system evaluates the nausea impact subscale and vomiting frequency score. Nausea impact subscale scoring will be rated by visual analogue scales (VAS) (0 = no impact to 10 = maximum impact). The VAS scores will be converted to 0-3 points via predefined thresholds. The Vomiting Frequency Score is categorized as follows: 0 for no episodes, 1 for 1-2 episodes, 2 for 3-5 episodes, and 3 for 6 or more episodes. The total score is calculated as the sum of the VAS-derived nausea impact score and the vomiting frequency score
Participant satisfaction with PONV management | At 6 hours, 24 hours, 48 hours, and 72 hours postoperatively
  Participant satisfaction will be also rated by visual analogue scales (VAS) (0 = very dissatisfied to 10 = most satisfied imaginable).
The use of rescue antiemetic drugs | During the 0-24 hours, 24-48 hours, and 48-72 hours postoperatively
  The use of rescue antiemetic drugs
The quality of postoperative recovery (QoR) | At 24 and 48 hours postoperatively, discharge, and 1 month postoperatively
  The quality of postoperative recovery (QoR) will be assessed by the 15-item quality of recovery scoring system [QoR-15]
The VAS scale | At 6 hours, 24 hours, 48 hours, and 72 hours postoperatively
  The VAS scale (0 = no pain to 10 = maximum pain)
Postoperative length of stay (LOS) | Within 1 month postoperatively
  Postoperative length of stay (LOS)
Safety outcomes | Within 1 month postoperatively
  Such as hypotension, bradycardia, hypertension, tachycardia, et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Luo, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- [Background] Rwei AY, Sherburne RT, Zurakowski D, Wang B, Kohane DS. Prolonged Duration Local Anesthesia Using Liposomal Bupivacaine Combined With Liposomal Dexamethasone and Dexmedetomidine. Anesth Analg. 2018 Apr;126(4):1170-1175. doi: 10.1213/ANE.0000000000002719. PMID 29239940
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162